CLINICAL TRIAL: NCT05497518
Title: The KidneyCARE (Community Access to Research Equity) Study: A National Registry for People With All Stages of Kidney Disease (Formerly National Kidney Foundation Patient Network)
Brief Title: The KidneyCARE (Community Access to Research Equity) Study
Status: Recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000053
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease; Dialysis; Kidney Transplant
Keywords: Chronic kidney disease; Dialysis; Kidney transplant; Patient registry; Hereditary nephropathy; Genetic kidney disease; Rare kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with chronic kidney disease: No interventions will be administered as part of this registry.
  Interventions: Other: Observational study - registry

INTERVENTIONS:
Other: Observational study - registry — The Study is a longitudinal observational cohort study that collaborates with health systems to obtain both electronic healthcare records (EHR) and patient-entered data. Eligible people with a diagnosis of chronic kidney disease at any stage, age 18 years and above, are identified through EHR data review, referral by a provider, or are recruited through the NKF's outreach campaign. Patients self-enroll into the online registry and share their experiences and health data through a secure portal where they can also find education, tips, and support. Research partners can view aggregate data through a collaboration portal.

SUMMARY:
For chronic kidney disease (CKD), there is a lack of unique and powerful platform for patient engagement, research studies and public health advocacy work. The National kidney Foundation (NKF) launched the first nationwide registry for people at all stages and types of CKD, including people on dialysis and kidney transplant recipients, called the KidneyCARE Study (kidneycarestudy.org). The KidneyCARE Study is a non-interventional research study which means participants will not have to take medications or do any additional tests to participate. They are simply asked to share some personal and health information, and their experiences with their disease through a secure portal. The Study also collaborates with health systems to obtain additional electronic health records (EHR) data. This unique combination of data collected will address the gap of individualized educational resources and will enhance clinical research, clinical care, and health policy decisions to be centered on the patient. The Study is all online and can be accessed any time of day at kidneycarestudy.org. Participation is voluntary and free.

DETAILED DESCRIPTION:
The KidneyCARE Study is a longitudinal prospective and retrospective observational cohort study of patient-entered data that collaborates with health systems to obtain additional electronic health records (EHR) data. The Study is approved by the Tufts Health Sciences Institutional Review Board, which serves as the IRB of record for all U.S. sites. The Study will start patient recruitment outside of the U.S. in 2022. The first international country will be Canada. The University of Manitoba, Winnipeg, MB, Canada is the Coordinating Site for all Canadian sites.

De-identified aggregate data is available for analysis to the NKF and the partners of the Study via analytic portals, dashboards, and/or subscription reports depending on contractual agreements. The individual site's data will be segregated from the rest of the registry, but the de-identified aggregate data can still be included in the overall registry's dashboard, reports, and analytics. Research proposals by partners and outside investigators that require advanced statistical analysis for publications in peer-reviewed journals, abstracts, and/or posters must be submitted and approved according to the Data Use and Publications policy. The Data Coordinating Center (DCC) conducts the statistical analyses for all approved research proposals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any stage of CKD, including kidney transplant recipients and patients on dialysis.
* Age 18 years and above.
* Willing to participate in the Study and complete the informed consent form and assent form (where applicable).
* Able to participate in this Study, which initially will be in English and then eventually expand to other languages.
* Patients affiliated with Geisinger Health System must have given their consent to Geisinger Health System IRB to be contacted for research projects.

Exclusion Criteria:

* Patient not diagnosed with CKD
* Age below 18 years
* Not willing to participate in the Study as well as unwilling to complete the informed consent form

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient recruitment targets two audiences: general public and closed systems. The general public is reached through a comprehensive outreach program that includes other NKF programs, local NKF field offices, participants from clinical trials for kidney disease treatments, referrals from other Network's participants, professional societies and patient advocacy groups, and a direct public relations campaign. The closed systems include health systems, academic medical centers, testing laboratories, or rare kidney disease groups. Here, patients will be recruited using the methods available at each organization (e.g., e-blasts, newsletters, provider/care manager recommendation, MyChart messages).
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2070-02-24 (Estimated); Study Completion 2070-02-24 (Estimated)

PRIMARY OUTCOMES:
Total number of enrolled participants | 5 years
  Reach 10,000 enrolled participants

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Willis, PhD, Study Director — National Kidney Foudnation
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inker LA, Ferre S, Baliker M, Barr A, Bonebrake L, Chang AR, Chaudhari J, Cooper K, Diamantidis CJ, Forfang D, Gillespie B, Gregoriou P, Gwadry-Sridhar F, Ladin K, Maxwell C, Mitchell KR, Murphy KP, Rakibuz-Zaman M, Rocco MV, Spry LA, Sharma A, Tangri N, Warfield C, Willis K; NKF Patient Network Governance Committees. A National Registry for People With All Stages of Kidney Disease: The National Kidney Foundation (NKF) Patient Network. Am J Kidney Dis. 2023 Feb;81(2):210-221.e1. doi: 10.1053/j.ajkd.2022.07.016. Epub 2022 Sep 30. PMID 36191726
- See also: Link for joining the first nationwide registry for people at all stages and types of kidney disease to transform kidney care and research together. — https://www.kidney.org/nkfpatientnetwork